CLINICAL TRIAL: NCT01201421
Title: Patient Satisfaction With Dental Restorations
Brief Title: DPBRN Patient Satisfaction With Dental Restorations
Status: Completed | Type: Observational
Sponsor: Dental Practice-Based Research Network (Network)
Collaborators: HealthPartners Institute (Other); Kaiser Permanente (Other); Permanente Dental Associates Group, Oregon (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Gregg H. Gilbert, DDS, MBA, Study Chair, University of Alabama at Birmingham
Other Study IDs: 118678; U01DE016747 (NIH)
Record Dates: First submitted 2010-09-13; First posted 2010-09-14 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Patient Satisfaction
Keywords: patient satisfaction; assessments; dental caries; dental materials
MeSH Terms: conditions — Patient Satisfaction; Dental Caries

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study was to administer two questionnaires. The first, a Dental Satisfaction Questionnaire to assess patient satisfaction with a restoration visit using patients recruited from practices participating in the Dental PBRN "Reasons for replacement or repair of dental restorations" study. The second questionnaire (completed by the practitioner) was a brief single page questionnaire to evaluate the patient visit.

DETAILED DESCRIPTION:
This study was to assess a comprehensive range of determinants of patient satisfaction following the restoration replacement or repair to study the relative contribution of each determinant towards overall patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* participants directly involved in this study were patients who sought dental treatment in the practitioner investigators' practices
* patient with replaced or repaired restorations placed in the treatment of permanent teeth who were also enrolled in the DPBRN "Reasons for replacement or repair of dental restorations"

Exclusion Criteria:

* children younger than 13 years of age were excluded from this study because of issues related to comprehension and validity of responses

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Practitioner investigators must have been enrolled in the DPBRN, completed the "Assessment of caries diagnosis & caries treatment" study; and do at least some restorative dentistry in their practices. The human subjects directly involved in this study were patients who had sought dental treatment in the DPBRN practitioners' practices.
Sampling Method: Non-Probability Sample
Enrollment: 5932 (Actual)
Dates: Start 2008-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregg H Gilbert, DDS, MBA, Study Chair — Dental Practice-Based Research Network; Joseph L Riley III, PhD, Principal Investigator — Dental Practice-Based Research Network
Locations (7):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Florida College of Dentistry, Gainesville, Florida
  - Health Partners Dental Group, Minneapolis, Minnesota
  - Health Partners Research Foundation, Minneapolis, Minnesota
  - Kaiser Permanente Center for Health Research, Portland, Oregon
  - Permanente Denrtal Associates, Portland, Oregon
- University of Copenhagen Royal Dental College, Copenhagen, Denmark